CLINICAL TRIAL: NCT03334448
Title: Bioequivalence Study Comparing the Pharmacokinetics and Glucodynamics of LY900014 U-200 Formulation With LY900014 U-100 Formulation in Healthy Subjects
Brief Title: A Study to Compare 2 Formulations of LY900014 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16636; I8B-MC-ITRQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2018-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY900014-U200 (Experimental): Single subcutaneous (SC) dose of 15 units (U) LY900014 U-200 in two of four study periods
  Interventions: Drug: LY900014-U200
- LY900014-U100 (Experimental): Single SC dose of 15 U LY900014 U-100 in two of four study periods
  Interventions: Drug: LY900014-U100

INTERVENTIONS:
Drug: LY900014-U200 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014-U200
Drug: LY900014-U100 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014-U100

SUMMARY:
The study involves a comparison of a LY900014 U-200 formulation with a LY900014 U-100 formulation. LY900014 is a type of fast acting insulin. Study participants will be administered LY900014 U-100 two times and LY900014 U-200 two times, over 4 study periods, by injection under the skin. Blood samples will be taken to compare how the body handles the study drugs and how they affect the blood sugar levels. Side effects and tolerability will be documented. The study will last about 4 weeks, not including screening and follow up. Screening is required within 28 days prior to the start of the study and follow up is required at least 2 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or a female (not pregnant and agreeable to take birth control measures until study completion)
* Have a body mass index (BMI) of 18 to 30 kilogram per square meter (kg/m²)
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Have veins suitable for easy blood collection and glucose solution infusion

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Had blood loss of more than 450 milliliters (mL) within the last 3 months
* Have a regular alcohol intake greater than 21 units/week (male), or 14 units/week (female)
* Smoke more than 10 cigarettes per day
* Are infected with hepatitis B or human immunodeficiency virus (HIV)
* Are taking illegal drugs

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Single subcutaneous (SC) dose sequences with 3 day washout between doses:
  A. LY900014 U-200 B. LY900014 U-100 C. LY900014 U-200 D. LY900014 U-100
- Sequence 2: Single subcutaneous (SC) dose sequences with 3 day washout between doses:
  A. LY900014 U-100 B. LY900014 U-200 C. LY900014 U-100 D. LY900014 U-200
- Sequence 3: Single subcutaneous (SC) dose sequences with 3 day washout between doses:
  A. LY900014 U-200 B. LY900014 U-100 C. LY900014 U-100 D. LY900014 U-200
- Sequence 4: Single subcutaneous (SC) dose sequences with 3 day washout between doses:
  A. LY900014 U-100 B. LY900014 U-200 C. LY900014 U-200 D. LY900014 U-100
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 12 | 13 | 12
Received at Least 1 Dose of Study Drug | 12 | 12 | 13 | 12
Completed | 12 | 12 | 13 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 12 | 13 | 12
Completed | 12 | 12 | 13 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 12 | 13 | 12
Received at Least 1 Dose of Study Drug | 12 | 12 | 13 | 12
Completed | 12 | 12 | 13 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 12 | 13 | 12
Completed | 12 | 11 | 13 | 12
Not Completed | 0 | 1 | 0 | 0
Not completed — Personal Reason | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 11 | 13 | 12
Received at Least 1 Dose of Study Drug | 12 | 11 | 13 | 12
Completed | 12 | 11 | 13 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 11 | 13 | 12
Completed | 12 | 11 | 13 | 11
Not Completed | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 11 | 13 | 11
Received at Least 1 Dose of Study Drug | 12 | 11 | 13 | 11
Completed | 12 | 11 | 13 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participant who received at least 1 dose of study drug.
Groups:
- Overall: All randomized participants who received at least 1 dose of study drug
Arm/Group | Overall
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 47
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 49
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 72.16 (10.97)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under Plasma Concentration Curve Zero to 10 Hours (AUC[0-10])
Description: Insulin Lispro AUC From Time Zero to 10 hours post dose (AUC[0-10h])
Time Frame: Predose, 5 minutes (mn), 10mn, 15mn, 20mn, 25mn, 30mn, 35mn, 40mn, 45 mn, 50mn, 55 mn, 60mn, 70mn,90mn,120mn,150mn,180mn, 240mn,300mn,360mn,320mn, 480mn, 540mn, and 600mn (10 hours)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours times picomols per milliliter
Groups:
- LY900014-U100: Single SC dose of LY900014 U-100 containing 15 units of insulin lispro in two of four study periods
- LY900014-U200: Single subcutaneous (SC) dose of LY900014 U-200 containing 15 units of insulin lispro (Humalog) in two of four study periods
Arm/Group | LY900014-U100 | LY900014-U200
Number analyzed (Participants) | 49 | 49
hours times picomols per milliliter | 1760 (19) | 1550 (42)
Statistical Analysis 1: Comparison: LY900014-U100 vs LY900014-U200; Test type: Superiority; Ratio of Geometric Least Square Means = 0.830, 90% CI 2-sided [0.818 to 0.957]

2. Secondary Outcome: Pharmacodynamics (PD): Total Amount of Glucose Infused (Gtot) Over Duration of Clamp for Each Treatment Arm
Description: Glucodynamics: Gtot is the total glucose infusion over the clamp duration (10 hours) and is used to measure the study drug action over time as measured by the euglycemic clamp (EC) procedure.
Time Frame: Predose, every minute from run-in and for the duration of the EC until up to 10 hours postdose
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per kilogram (mg/kg)
Arm/Group | LY900014-U100 | LY900014-U200
Number analyzed (Participants) | 49 | 49
milligrams per kilogram (mg/kg) | 1500 (47) | 1410 (55)
Statistical Analysis 1: Comparison: LY900014-U100 vs LY900014-U200; Test type: Superiority; Ration of Lease Square Means = 0.97, 90% CI 2-sided [0.83 to 1.09]

ADVERSE EVENTS:
Time Frame: Up to 15 months
Description: All participants who received at least 1 dose of study drug.
Arm/Group | LY900014-U100 | LY900014-U200
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 32/49 | 35/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014-U100 (N=49) | LY900014-U200 (N=49)
Catheter site bruise (General disorders) | 6 (8) | 6 (9)
Catheter site pain (General disorders) | 4 (5) | 2 (2)
Catheter site swelling (General disorders) | 6 (9) | 2 (3)
Infusion site bruising (General disorders) | 3 (3) | 6 (6)
Infusion site pain (General disorders) | 6 (6) | 10 (12)
Infusion site swelling (General disorders) | 5 (6) | 4 (4)
Injection site reaction (General disorders) | 23 (30) | 16 (18)
Pyrexia (General disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT03334448/SAP_000.pdf
  • Study Protocol (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03334448/Prot_001.pdf